CLINICAL TRIAL: NCT02662959
Title: A Phase II Study of Irinotecan as Single Agent in the Third Line Treatment of Unresectable or Metastatic Gastric Cancer.
Brief Title: Irinotecan as 3rd Line Therapy in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Med Onc-G 01
Record Dates: First submitted 2015-04-23; First posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-11

CONDITIONS: Stomach Neoplasms
Keywords: Chemotherapy, metastatic gastric cancer, irinotecan
MeSH Terms: conditions — Stomach Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irinotecan (Experimental): In the experimental arm, patients receive single agent of irinotecan as third line treatment in metastatic gastric cancer.
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — 180 mg/m2, IV (in the vein) on day 1 of each 14 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.

SUMMARY:
Gastric cancer is the leading cause of cancer death in China. Most patients are unresectable or metastatic disease at the time of diagnosis. Systemic therapy was required for the patients with advanced stage. Platinum combined with fluoropyrimidines always were considered as first line treatment. After failure of initial therapy, single agent of taxanes was used as second line treatment. However, there is no relative standard chemotherapeutic regimen in the third therapy except oral anti-angiogenesis drug-Apatinib. So this study was designed to explore the role of single agent with irinotecan as third line treatment in patients with metastatic gastric cancer in China.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic adenocarcinoma of the stomach
* Have failed for 2 lines of chemotherapy
* Life expectancy of more than 3 months
* ECOG performance scale ≤ 2
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* Duration from the last therapy is more than 6 weeks for nitroso or mitomycin
* More than 4 weeks for operation or radiotherapy
* More than 4 weeks for cytotoxic agents or growth inhibitors
* Adequate hepatic, renal, heart, and hematologic functions (platelets > 100 × 109/L, neutrophil > 1.5× 109/L, serum creatinine ≤ 1×upper limit of normal(ULN), total bilirubin within 1× ULN, and serum transaminase≤2.5×the ULN).
* Exclusion of pregnant or lactating women

Exclusion Criteria:

* Previously receiving irinotecan treatment
* Participated other clinical trials within 4 weeks
* Known Gilbert Syndrome or other biliary tract obstructive disease
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Evidence of CNS metastasis
* Intercurrence with one of the following: hypertension, coronary artery disease, arrhythmia and heart failure
* Receiving the therapy of thrombolysis or anticoagulation
* Disability of serious uncontrolled intercurrence infection.
* Uncontrolled pleural effusion and ascites

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1 year
  From the day enrolled in the study to death

SECONDARY OUTCOMES:
Progression free survival | 6 month
Objective Response Rate | 8 weeks
  evaluated by RECIST 1.1
Number of Adverse Events | Participants will be followed for the duration of treatment interval, an expected average of two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yu N, Huang S, Zhang Z, Huang M, Wang Y, Zhang W, Zhang X, Zhu X, Sheng X, Yu K, Chen Z, Guo W. A prospective phase II single-arm study and predictive factor analysis of irinotecan as third-line treatment in patients with metastatic gastric cancer. Ther Adv Med Oncol. 2024 Feb 28;16:17588359241229433. doi: 10.1177/17588359241229433. eCollection 2024. PMID 38425987